CLINICAL TRIAL: NCT05517070
Title: Association of Vitamin D Deficiency, Sarcopenia, Body Composition, Osteoporosis and Hemophilic Arthropathy in the Patients With Hemophilia
Brief Title: Vitamin D Deficiency and Body Composition in the Patients With Hemophilia
Status: Completed | Type: Observational
Sponsor: Tsung-Ying Li (Other)
Responsible Party: Sponsor-Investigator, Tsung-Ying Li, Attending Physician, Tri-Service General Hospital
Organization: Tri-Service General Hospital (Other)
Other Study IDs: 1-108-05-001
Record Dates: First submitted 2022-08-24; First posted 2022-08-26 (Actual); Last update posted 2024-08-13 (Actual); Status verified 2024-08

CONDITIONS: Vitamin D Deficiency; Sarcopenia; Osteoporosis; Body Composition; Hemophilic Arthropathy; Hemophilia
MeSH Terms: conditions — Vitamin D Deficiency; Sarcopenia; Osteoporosis; Hemophilia A

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Hemophilia Group: Hemophilia adult patients
- Control Group: Healthy adult subjects

SUMMARY:
Hemophilia is associated with osteoporosis and increased prevalence of low bone mineral density (BMD). Many clinical risk factors have been reported, such as hemophilic arthropathy, reduced physical activity, decreased sun exposure, hepatitis C virus infections, vitamin D deficiency, and low body mass index (BMI). There is no data on the prevalence of vitamin D deficiency and low BMD in hemophilia patients in Taiwan or Asia. To the best of our knowledge, no previous studies have reported the prevalence of sarcopenia and correlation with osteoporosis in hemophilia adult patients. The purpose of this study will evaluate the prevalence of vitamin D deficiency, low BMD, sarcopenia and body composition in a cohort of patients with hemophilia in Taiwan.

DETAILED DESCRIPTION:
Hemophilia is associated with osteoporosis and increased prevalence of low bone mineral density (BMD). Soucek et al. reported sarcopenia and low trabecular BMD at the radius in the boys with hemophilia by CT.The severity of hemophilic arthropathy associated with lower BMD, muscle atrophy and obesity has been shown by some studies.

This is a single-center, cross-sectional, observational study. All participants will sign informed consent that fully disclosed the risks and benefits of study participation. The study will be performed at the Hemophilia Care and Research Center. Sixty adult patients (age ≥ 20) with hemophilia and 20 healthy subjects will be enrolled for scanning of the lean tissue, appendicular skeletal muscle mass (ASM), fat mass, lumbar spine and hip BMD by dual-energy X-ray absorptiometry (DXA) and assess serum vitamin D level. We will collect other clinically relevant information, including age, body mass index (BMI), hemophilia type and severity, inhibitor titer, Pettersson score by x-ray, HJHS, handgrip strength, history of HCV or HIV infection and history of fracture.

ELIGIBILITY:
Inclusion Criteria:

* Hemophilia patients

Exclusion Criteria:

* Severe diseases affecting bone metabolism (such as primary hyperparathyroidism, hypogonadism),
* History of total hip arthroplasty
* History of instrumentation in lumbar spine

Min Age: 20 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: 60 hemophilia patients and 20 healthy subjects
Sampling Method: Non-Probability Sample
Enrollment: 80 (Actual)
Dates: Start 2021-01-01 (Actual); Primary Completion 2023-12-31 (Actual); Study Completion 2023-12-31 (Actual)

PRIMARY OUTCOMES:
Vitamin D | one day
  serum vitamin D

SECONDARY OUTCOMES:
Bone marrow density | one day
  Bone marrow density of lumbar spine and bilateral hip by dual X-ray absorptiometry (DXA)
Body composition | one day
  using whole-body DXA (GE Lunar iDXA, GE Healthcare Lunar, Madison, Wisconsin, U.S.A.)
Pettersson score | one day
  Bilateral shoulder, elbow, hip, knee, ankle joints score by x-ray. The Pettersson score ranges from 0 (normal) to 13 (most severe) and is according to the following eight radiographic features of joints: osteoporosis, osteophytes, narrowing of joint space, subchondral irregularity, subchondral cyst formation, erosion of joint margins, and bone remodelling.
Hemophilia Joint Health Score | one day
  Functional and structured score of bilateral elbow, knee and ankle. The score for each joint is the sum of several elements including swelling (0-3), duration of swelling (0-1), muscle atrophy (0-2), crepitus of motion (0-2), flexion loss and extension loss (0-6), joint pain (0-2) and strength (0-4). A score of 20 may indicate the most severe damage/impairment in the evaluated joint and a score of zero corresponds to no identifiable joint impairment.
Handgrip strength | one day
  Handgrip strength (kg) will be measured using the same standard calibrated hand dynamometers (Baseline® Hand Dynamometer - Digital LCD Gauge, Fabrication Enterprises Inc. White plains, New York, USA). We will calculate the mean of three maximal grip-strength measurement in each hand.

CONTACTS AND LOCATIONS:
Overall Officials: Tsung Ying Li, Dr, Principal Investigator — No.325,Sec.2, Cheng-Kung Rd. Neihu 11490, Taipei, Taiwan, R.O.C
Locations (1):
- Hemophilia care and research center, Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: No